CLINICAL TRIAL: NCT04173481
Title: Effects of ROOD's Sensory Motor Training Along With Constraint Induced Movement Therapy in Sub-acute Stroke
Brief Title: ROOD's Sensory Motor Training in Sub-acute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RiphahIUAroosaTariq
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Stroke
Keywords: Stroke; Proprioceptive Neuromuscular Facility; Hemiplegia; Neurorehabilitation; Neural Plasticity
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rood's Group (Experimental): Rood's sensory motor training along with CIMT
  Interventions: Other: Rood's Group
- Conventional Physical Therapy Group (Active Comparator): Conventional Physical Therapy including Proprioceptive Neuromuscular Facilitation technique.
  Interventions: Other: Conventional Physical Therapy Group

INTERVENTIONS:
Other: Rood's Group — ROOD'S sensory motor training
  Brushing & strokings 3-5 strokings after 30sec, joint compressions and slow stretch 10 rep of 3 sets on alternative days for consecutive 6 weeks CIMT training
  Writing, combing hairs and using spoon activity 1 hour training concentrated on affected limb along with restraint of non affected limb by cotton sling under supervision of therapist and 5 hours training in home plan 3 times a week on alternative days for consecutive 6 weeks along with conventional physical therapy.
  Arms: Rood's Group
Other: Conventional Physical Therapy Group — Conventional training Proprioceptive neuromuscular facilitations (PNF) Combination of Isotonics technique 10 rep 3 sets 10 sec hold on alternative days for consecutive 6 weeks Stretching's 10 rep 3 sets on alternative days for consecutive 6 weeks Joint approximation 10 rep of 3 sets on alternative days for 6 weeks
  Arms: Conventional Physical Therapy Group

SUMMARY:
The aim of this randomized controlled trial is to determine the effects of ROOD's sensory motor training along with Constraint Induced Movement Therapy (CIMT) in sub-acute stroke. Two randomized groups of patients with stroke were treated with conservative physical therapy and the experimental group was given ROOD's SMT and CIMT in conjunction with conservative rehabilitation. Both, male and female patients meeting the inclusion criteria were included. Patients having other neurological disease, chronic disease, not compatible being participates in CIMT or with any surgical intervention were excluded.

DETAILED DESCRIPTION:
The study is aimed at determining the effects of ROOD's sensory motor training along with constraint induced movement therapy in sub-acute stroke and is being conducted in National Institute of Rehabilitation Medicine Islamabad and Pakistan Railway General Hospital, Rawalpindi (Feb 2019-July 2019). Sample size of the study is 36 patients, 36 were included in the study on the basis of inclusion criteria, 18 for each group. Patients were allocated randomly and equally in each group. Similar conservative rehabilitation protocol was designed for both control and experimental group except for experimental group had ROOD's sensory motor training and CIMT training. Patients were examined at 1st visit before administration of any treatment and at 6th week which was also the last one (after completing 6 weeks sessions at alternate days). Baseline evaluation for demographics and assessment was taken. Fugyl-meyer assessment scale(FMA) and Wolf motor function test(WMFT) as measuring tools were used for first and 6th week assessment. 29 patients completed the study while 4 patient from control group and 3 patients from experiment group were lost to follow up and were considered drop outs.

ELIGIBILITY:
Inclusion Criteria:

* Right & Left hemiplegia
* Ischemic & Hemorrhagic stroke
* Compatible with being participate in CIMT i.e. 10ºwrist extension,10ºany two fingers extension,10ºthumb abduction
* Duration of stroke between 6 weeks to 6 months

Exclusion Criteria:

* Not compatible with being participate in CIMT
* Any other neurological disease e.g. Parkinson's disease, brain tumors
* Chronic disease e.g. Ischemic Heart Disease, tumors, Diabetes Mellitus
* Behaviors issues, not willing to participate
* Surgical intervention that hinders treatment and assessment
* Not well oriented to follow designed motor task

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Wolf Motor Function Test | 6 weeks
  Changes from the baseline, Wolf motor function test is a test of motor ability that is use to evaluate the speed and coordination.
  Total of 17 tasks performed by the patient.
  Scoring:
  The items are rated on a 6-point scale as 0-6.
Fugyl-meyer motor assessment scale | 6 weeks
  Changes from the baseline, Fugyl-meyer assessment scale is use to assess voluntary movements, reflex activity, grasping and coordination of affected limb in stroke. FMA upper extremity portion contain 33 tasks with a scale 0 to 2 with maximum scoring of 66.

CONTACTS AND LOCATIONS:
Overall Officials: Mir Arif Hussain, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sacco RL, Kasner SE, Broderick JP, Caplan LR, Connors JJ, Culebras A, Elkind MS, George MG, Hamdan AD, Higashida RT, Hoh BL, Janis LS, Kase CS, Kleindorfer DO, Lee JM, Moseley ME, Peterson ED, Turan TN, Valderrama AL, Vinters HV; American Heart Association Stroke Council, Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular and Stroke Nursing; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Council on Nutrition, Physical Activity and Metabolism. An updated definition of stroke for the 21st century: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Jul;44(7):2064-89. doi: 10.1161/STR.0b013e318296aeca. Epub 2013 May 7. PMID 23652265
- [Background] Redon J, Olsen MH, Cooper RS, Zurriaga O, Martinez-Beneito MA, Laurent S, Cifkova R, Coca A, Mancia G. Stroke mortality and trends from 1990 to 2006 in 39 countries from Europe and Central Asia: implications for control of high blood pressure. Eur Heart J. 2011 Jun;32(11):1424-31. doi: 10.1093/eurheartj/ehr045. Epub 2011 Apr 12. PMID 21487117
- [Background] Umar M, Badshah M, Baig MS. Frequency of Dystonia Among Post Stroke Patients in Pakistan. Annals of PIMS ISSN. 2016;1815:2287.
- [Background] Langhorne P, Bernhardt J, Kwakkel G. Stroke rehabilitation. Lancet. 2011 May 14;377(9778):1693-702. doi: 10.1016/S0140-6736(11)60325-5. PMID 21571152
- [Background] Doyle S, Bennett S, Fasoli SE, McKenna KT. Interventions for sensory impairment in the upper limb after stroke. Cochrane Database Syst Rev. 2010 Jun 16;2010(6):CD006331. doi: 10.1002/14651858.CD006331.pub2. PMID 20556766
- [Background] Lang CE, Bland MD, Bailey RR, Schaefer SY, Birkenmeier RL. Assessment of upper extremity impairment, function, and activity after stroke: foundations for clinical decision making. J Hand Ther. 2013 Apr-Jun;26(2):104-14;quiz 115. doi: 10.1016/j.jht.2012.06.005. Epub 2012 Sep 10. PMID 22975740
- [Background] Sawaki L, Butler AJ, Leng X, Wassenaar PA, Mohammad YM, Blanton S, Sathian K, Nichols-Larsen DS, Wolf SL, Good DC, Wittenberg GF. Constraint-induced movement therapy results in increased motor map area in subjects 3 to 9 months after stroke. Neurorehabil Neural Repair. 2008 Sep-Oct;22(5):505-13. doi: 10.1177/1545968308317531. PMID 18780885
- [Background] Kwakkel G, Veerbeek JM, van Wegen EE, Wolf SL. Constraint-induced movement therapy after stroke. Lancet Neurol. 2015 Feb;14(2):224-34. doi: 10.1016/S1474-4422(14)70160-7. PMID 25772900
- [Background] Shi YX, Tian JH, Yang KH, Zhao Y. Modified constraint-induced movement therapy versus traditional rehabilitation in patients with upper-extremity dysfunction after stroke: a systematic review and meta-analysis. Arch Phys Med Rehabil. 2011 Jun;92(6):972-82. doi: 10.1016/j.apmr.2010.12.036. PMID 21621674
- [Background] Schriner M, Thome J, Carrier M. Rehabilitation of the upper extremity after stroke: current practice as a guide for curriculum. The Open Journal of Occupational Therapy. 2014;2(1):6.
- [Background] Pollock A, Baer G, Campbell P, Choo PL, Forster A, Morris J, Pomeroy VM, Langhorne P. Physical rehabilitation approaches for the recovery of function and mobility following stroke. Cochrane Database Syst Rev. 2014 Apr 22;2014(4):CD001920. doi: 10.1002/14651858.CD001920.pub3. PMID 24756870
- [Background] Nijland R, van Wegen E, Verbunt J, van Wijk R, van Kordelaar J, Kwakkel G. A comparison of two validated tests for upper limb function after stroke: The Wolf Motor Function Test and the Action Research Arm Test. J Rehabil Med. 2010 Jul;42(7):694-6. doi: 10.2340/16501977-0560. PMID 20603702
- [Background] Sullivan KJ, Tilson JK, Cen SY, Rose DK, Hershberg J, Correa A, Gallichio J, McLeod M, Moore C, Wu SS, Duncan PW. Fugl-Meyer assessment of sensorimotor function after stroke: standardized training procedure for clinical practice and clinical trials. Stroke. 2011 Feb;42(2):427-32. doi: 10.1161/STROKEAHA.110.592766. Epub 2010 Dec 16. PMID 21164120
- [Background] Beekhuizen KS, Field-Fote EC. Sensory stimulation augments the effects of massed practice training in persons with tetraplegia. Arch Phys Med Rehabil. 2008 Apr;89(4):602-8. doi: 10.1016/j.apmr.2007.11.021. PMID 18373988